CLINICAL TRIAL: NCT06440668
Title: Management of Chronic Non-Cancer Pain With Non-Pharmacological Therapies: Randomized Clinical Trial.
Brief Title: Management of Chronic Non-Cancer Pain With Non-Pharmacological Therapies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Juan de Dios del Aljarafe de Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-2024
Record Dates: First submitted 2024-05-14; First posted 2024-06-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain Syndrome; Sensitization, Central; Quality of Life; Patient Empowerment
Keywords: Chronic Pain Syndrome; Sensitization, Central; Quality of Life; Patient Empowerment
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial
Who Masked: Investigator
Masking Description: The statistician who analyse the data is unaware of the group to which each patient belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop (Experimental): Psychoeducational and self-care training, pain management, and emotional control, conducted in groups and aimed at patients with non-cancer chronic pain. Therapies applied: relaxation, meditation, cognitive-behavioral therapy, acceptance and commitment therapy, coaching, healthy eating, physical exercise, improving self-esteem, forgiveness technique. This group starts and successfully completes the workshop. A patient is considered to have successfully completed if they: Attend at least 4 out of the 5 sessions; complete all the initial documentation, at the end of the workshop, and at the 3-month mark; perform daily tracking of the 3 mandatory activities throughout the duration of the workshop.
  Interventions: Behavioral: Chronic Pain Management Workshop with Non-Pharmacological Therapies
- Traditional treatment (No Intervention): This group meets the inclusion criteria but does not participate in the workshop. They complete all documentation at the beginning, at one month, and at three months. These patients will continue with the usual treatment prescribed by their doctor.

INTERVENTIONS:
Behavioral: Chronic Pain Management Workshop with Non-Pharmacological Therapies — 1st Session: Welcome. Expectations. Pathophysiological mechanism of pain. Influence of emotions on pain intensity. Activities: My limiting beliefs; Affirmations in front of the mirror; Mental analgesia. / 2nd: Pain and its impact on the patient's life. Forgiveness and self-forgiveness. Ho'oponopono technique. Self-esteem. Activities: Labels that limit us; Reading "When I Loved Myself for Real"; Self-healing meditation; Life purpose. / 3rd: Tips to slow down aging. Promotion of healthy habits; Metta meditation; Motivation for change. / 4th: Active participation in my own healing. How to face illness. Creative visualization. Activity:Energy wheel. / 5th: Review of the tools. Resolving doubts. Workshop evaluation and scales. Guide with the tools presented. Activities: Final farewell. / At the end of each session, the homework assignments are explained, and at the beginning of the next, they are reviewed. Sessions 2, 3, 4 5: Experience of a previous workshop patient.
  Arms: Workshop

SUMMARY:
A randomized controlled clinical trial will be conducted, involving a psychoeducational activity as the intervention. There will be a control group of patients with non-cancer chronic pain who will continue their usual treatment.

The trial will end after 3 months. Pain, well-being, medication management, mood, self-esteem, and quality of life will be compared just before starting the workshop with the status at the end of the workshop (one month later) to assess the immediate effect, and three months later to evaluate the medium-term effect. These measurements will be taken in both the control and intervention groups.

Additionally, for the intervention group, a follow-up will be conducted six months after the workshop ends to assess the long-term effect duration.

This study does not allow blinding of patients or professionals conducting the intervention, but the person analyzing the data to compare the effect produced in the control and intervention groups will be blinded. Therefore, it is an observer-blind evaluation.

DETAILED DESCRIPTION:
Intervention Group: Workshop. This group starts and completes the workshop (attend at least 4 out of the 5 sessions). Complete all the initial documentation, at the end of the workshop, and at the 3-month mark. Perform daily tracking of the 3 mandatory activities throughout the duration of the workshop.

Control Group: Traditional treatment. This group meets the inclusion criteria but does not participate in the workshop. They complete all documentation at the beginning, at one month, and at three months. These patients will continue with the usual treatment prescribed by their doctor.

Intervention: Chronic Pain Management Workshop with Non-Pharmacological Therapies. Psychoeducational and self-care training, pain management, and emotional control, conducted in groups and aimed at patients with non-cancer chronic pain.

Workshop Methodology and Facilities: It will take place at HSJDA over 5 afternoons, with each session lasting 3.5 hours. Sessions will be held once a week for 5 consecutive weeks.

The sessions will include oral presentations supported by PowerPoint, videos, activities to be performed in the classroom by the patients to apply different techniques, testimonies from individuals known for personal overcoming, experiences from patients of previous workshops, and the application of the explained tools.

In the first session, a WhatsApp group will be created with the participants of each workshop, coordinated by a volunteer patient, who will directly contact the workshop director. The director will send reinforcement information from the workshop sessions, such as videos and songs, through this group.

Patients can ask questions via the group, which will be directed from the patient coordinator to the workshop director for resolution. They can also report any issues regarding attendance to a session.

This group will remain active for up to 6 months to serve as reinforcement and a support group for the patients. At the end of each session, patients will be given some homework for the week, as well as a tracking sheet to record 3 activities they must perform daily and an assessment of pain control using the main technique (to be filled out daily until the workshop ends).

In the last session, there will be a review of all the tools presented in previous sessions, questions will be answered, and patients will evaluate the workshop (satisfaction, most useful aspects, etc.), as well as its impact on pain control and other aspects (quality of life, self-esteem, mood, etc.). They can also provide suggestions for improvement and free-text comments.

At the end of the workshop, patients will receive a guide reinforcing what was explained in the workshop so they can continue applying the tools and recommendations after the workshop ends.

Patient Recruitment: Patients will be referred by healthcare professionals from the following services or areas: Rehabilitation, Traumatology, Internal Medicine, Gynecology, etc. Primary Care: Health Centers in the Aljarafe Area belonging to the Aljarafe-Sevilla Norte Health District. Associations of patients with conditions associated with non-cancer chronic pain.

Sample Selection: Each referred patient will be interviewed by phone by the workshop director to confirm they meet the inclusion criteria. If they do, they will be informed about the workshop, invited to participate in the study, and if they accept, they will be sent the information sheet and informed consent via email, to be returned signed by email.

All those who accept will be added to the list of workshop candidate patients registered in Excel. Participants will be assigned to each group (control and intervention) using the Excel "RAND" function, which assigns a random number to each patient, then sorted from smallest to largest, with the first half forming the control group and the other half forming the intervention group.

Sample Size: Each workshop will include a maximum of 20 patients. A 20% dropout rate is expected (patients missing two or more sessions), so approximately 16 patients are expected to complete each workshop. Using G*POWER software, the sample size calculation was performed using an independent samples t-test to compare means of two groups (control and experimental), considering a significance level of 0.05, power of 0.80, and an effect size of 0.5 (conservative size), resulting in a sample size of 128 patients (64 in each group).

Workshops will be conducted until the required sample size is recruited. Considering a 20% dropout rate, 4 workshops will be needed, recruiting 80 patients (20 per workshop), expecting 80% to complete the workshops, resulting in 64 patients, meeting the minimum sample size required.

Workshop Follow-up: Both control and experimental groups will undergo 3 measurements: initial, one month (workshop end), and three months, completing the clinical trial. Additionally, the experimental group will have a follow-up one month after completion (two months from the start), presenting group results (anonymized) and a brief personalized report of their results. Another follow-up will occur at six months to assess if the workshop effect persists long-term, with the scales administered again.

Statistical Analysis: With the documentation collected at the beginning of the study, the random allocation will be ratified, checking the comparability of all variables that may influence the final outcome. Descriptive statistics will be performed in each group:

Continuous quantitative variables: mean and SD (if they follow a normal distribution); median and quartiles (if they do not follow a normal distribution). Categorical variables: Absolute and relative frequencies (%). The normality of the variables will be checked with the Kolmogorov-Smirnov test.

95% confidence intervals will be calculated for means and percentages. At the end of the study, an intention-to-treat analysis will be performed. The Statistical Package for Social Sciences (SPSS) Version 27.0 will be used.

To compare the main and secondary dependent variables between the control and intervention groups, hypothesis testing will be performed: Student's t-test and ANOVA (for quantitative variables that follow a normal distribution), Mann-Whitney U and Kruskal-Wallis (for those with a non-normal distribution) when comparing 2 or more groups, respectively.

To compare related variables (before and after) both within the control group and within the intervention group, paired t-tests will be used for normally distributed data, and the Wilcoxon test for non-normally distributed data.

The correlation between outcome variables will also be assessed using Pearson's or Spearman's correlation coefficient, depending on whether the variables compared follow a normal distribution or not. The normality of quantitative variables will be checked using the Kolmogorov-Smirnov test.

For qualitative variables, the Chi-square test or Fisher's test (if expected frequencies are low) will be used to compare independent variables, and the McNemar test to compare related variables.

Finally, a multivariate analysis will be conducted to develop an explanatory model with the main variables that influence the outcomes. The Odds Ratio of the associations with their confidence intervals will be calculated.

Bioethical considerations. This project, has received favorable approval from the Research Ethics Committee of the University Hospitals Virgen Macarena and Virgen del Rocío at its meeting on 20/07/2023, under record CEI_07/2023. Internal Code: 1181-N-23. Researchers involved in this project will ensure compliance with current regulations and legislation governing research involving human subjects (Declaration of Helsinki and its update in Fortaleza (Brazil), Oviedo Declaration, Good Clinical Practice Guide of the ICH -CPMP/ICH/135/95-, Law 41/2002 of November 14, regulating patient autonomy, Law 14/2007 of July 3, on biomedical research).

Individuals participating in this project must have provided written consent once they have been adequately informed and their questions have been addressed. Researchers will ensure the anonymity and the confidentiality of participants' data (recommendations of REGULATION (EU) 2016/679 OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of April 27, 2016; Directive 95/46/EC and Organic Law 3/2018, of December 5, on Personal Data Protection and guarantee of digital rights. Two databases (DB) will be worked with and kept in different files. In DB-1, the NID (patient identification number) will be related to personal data. The NID is a unique number for each patient. In DB-2, the NID will be related to patients' clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older,
* Residing in the areas served by HSJDA,
* With non-cancer chronic pain already diagnosed and treated for at least 6 months but not relieved by the usual treatment,
* Who have explicitly and in writing expressed their desire to participate in the workshops and the study through the Informed Consent document,
* And who complete the initial documentation necessary for their evaluation.

Exclusion Criteria:

* Patients in the diagnostic phase,
* Patients with pain exclusively associated with cancer pathology,
* Patients with a life expectancy of less than one year,
* Patients with severe cognitive or mental illnesses that prevent them from understanding both the content of the workshops and the measurement instruments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain last week | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Pain measured with the "visual analogue scale" (scale: 0-10)
Analgesic regimen | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  self-assessment at the end of the workshop on whether they have replaced a higher-tier analgesic with a lower one, decreased the dosage, reduced the frequency, or stopped taking analgesics or anxiolytics/antidepressants.
Well-being | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Numerical visual scale from 0 (minimum) to 10 (maximum). Higher scores indicate greater well-being.
Self-esteem | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Rosenberg Self-esteem Scale, ranging from 9 (minimum) to 36 (maximum).Higher scores indicate greater Self-esteem
Anxiety and Depression | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Hospital Anxiety and Depression Scale (HADS). It consists of 14 items with two subscales (anxiety and depression), each with scores from 0 to 3. Cut-off points: <8 normal, 8-10 possible cases, and >10 for cases in both subscales.
Resilience | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Brief Resilience Scale (BRS). Scale from 6 (minimum) to 30 (maximum). Higher scores indicate greater resilience.
Health-related quality of life | 4 measurements: The scale will be administered just before starting the workshop, at the end (last day of the workshop, after 4 weeks), at 3 months, and at 6 months (this only in the intervention group).
  Measured with the EuroQol-5D questionnaire. Scale from 0 to 1 (maximum) (with the possibility of negative values). Higher scores indicate greater health-related quality of life.
Number of emergency episodes and outpatient visits | 3 measurements: The scale will be administered just before starting the workshop, at 3 months, and at 6 months (this only in the intervention group).
  The number of emergency episodes and outpatient visits for pain or associated symptoms (anxiety, depression, insomnia) will be quantified, both in primary care (at their health center) and hospitalized.

SECONDARY OUTCOMES:
Satisfaction with the workshop | 1 measurement: The scale will be administered just at the end (last day of the workshop, after 4 weeks) (this only in the intervention group).
  Satisfaction with the workshop: Clarity of the presented content; Appropriateness of the exercises and activities performed; Usefulness of the workshop for managing my pain; Usefulness of the workshop for managing my illness; To what extent would you recommend this workshop?; Overall satisfaction. Suggestions for improvement are also collected. Scale from 0 to 10.
Improving habits | 2 measurements: In the 3rd session and just at the end (last day of the workshop, after 4 weeks) (this only in the intervention group).
  In the 3rd session, we work on a self-assessment of certain habits (nutrition, physical exercise, relaxation/meditation, "me time") and ask participants to choose one or two to improve and make the change. At the end of the workshop, we ask them if they have made any habit changes and what those changes were, through the self-assessment questionnaire they complete at the end of the workshop. This is measured as Yes/No.

CONTACTS AND LOCATIONS:
Locations (1):
- María Victoria RUIZ ROMERO, Bollullos de la Mitación, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No
We will not be shared with other researchers individual participant data.

REFERENCES:
- [Background] Ruiz Romero MV, Lobato Parra E, Porrua Del Saz A, Martinez Monrobe MB, Pereira Delgado CM, Gomez Hernandez MB. [Management of chronic non-oncologic pain by multicomponent programs using non-pharmacologic therapies: A systematic review of the literature]. J Healthc Qual Res. 2024 May-Jun;39(3):168-187. doi: 10.1016/j.jhqr.2024.02.004. Epub 2024 Mar 30. Spanish. PMID 38556371
- [Background] Ruiz Romer MV, Porrua Del Saz A, Gomez Hernandez MB, Lobato Parra E, Soler Jimenez A, Pereira Delgado C. [Impact of a multicomponent program with nonpharmacological therapies for patients with chronic pain]. J Healthc Qual Res. 2024 Mar-Apr;39(2):109-119. doi: 10.1016/j.jhqr.2024.01.005. Epub 2024 Feb 23. Spanish. PMID 38402091
- [Background] Ruiz Romero MV, Lopez Tarrida AC, Porrua Del Saz A, Gomez Hernandez MB, Martinez Monrobe MB, Sanchez Villar E, Cruz Valero C, Pereira Delgado C. [Efectividad de una intervencion multimodal para la mejora de la atencion al dolor cronico.]. Rev Esp Salud Publica. 2023 Sep 6;97:e202309071. Spanish. PMID 37921370
- [Background] Ruiz-Romero MV, Guerra-Martin MD, Alvarez-Tellado L, Sanchez-Villar E, Arroyo-Rodriguez A, Sanchez-Gutierrez MC. [Non-drug treatments for chronic non-malignant pain]. An Sist Sanit Navar. 2022 Aug 30;45(2):e1011. doi: 10.23938/ASSN.1011. No abstract available. Spanish. PMID 36040235